CLINICAL TRIAL: NCT00629174
Title: Randomized, Controlled Study About the Effects of an Exercise Program and Mental Activity on the Age-Associated Impairment of Cognitive Function
Brief Title: Prevention of the Age-Related Cognitive Impairment by Exercise and Mental Activity - Berlin Bleibt Fit
Acronym: BBF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other); Gertrude and Hugo Adler Foundation (Other)
Responsible Party: Prof. Isabella Heuser, Prof. Friedel Reischies, Dr. Fernando C. Dimeo, Charité - Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 28_12_2005
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Cognition; Mood
Keywords: Cognitive function; Elderly; Exercise; Mental activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Exercise
  Interventions: Behavioral: Exercise
- 2 (Experimental): Mental training (computer lessons)
  Interventions: Behavioral: Mental activity
- 3 (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — Endurance and resistence training, 90 minutes, 3 times weekly
  Arms: 1
Behavioral: Mental activity — Participation at computer lessons, 3 times weekly, 90 minutes each
  Arms: 2

SUMMARY:
The trial will evaluate the effects of frequent exercise and increased mental activity on the age-related impairment of cognitive function in elderly women. Furthermore, we will assess the effects of exercise and mental activity on the mood, physical performance and mental status of participants. We will also search for genetic factors which may be responsible of the observed outcomes.

DETAILED DESCRIPTION:
Two-hundred and fifty-two women older than 70 years will be randomize to one of three groups. The first (exercise) will participate at an exercise program three times weekly for 90 minutes. The training will consist of an endurance and resistance training and will be carried out in a group. Participants in the second group (mental training) will take computer lessons, three times weekly for 90 minutes. Both interventions will be carried out for 26 weeks. Participants in the third group (control) will not participate at an structured intervention.

ELIGIBILITY:
Inclusion Criteria:

* All healthy women older than 70 years with sufficient knowledge of German can participate.

Exclusion Criteria:

* Chronic mental disorders
* Chronic neurological, cardiological, pulmonary or renal diseases.
* Severe osteoarthritis
* Disorders which can be aggravated by exercise (arterial hypertension, coronary heart disease, COLD).
* Cancer in current therapy
* Treatment with glucocorticoids or cytostatic drugs.
* Patients who received an organ transplantation
* Exercise-induced osteoarticular pain

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of cognitive and physical performance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Heuser, Professor, Study Chair — Charite University, Berlin, Germany; Fernando C Dimeo, PhD, Study Chair — Charite University, Berlin, Germany; Friedel Reischies, Professor, Study Chair — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Section Sports Medicine, Charité - Universitätsmedizin Berlin, Berlin
  - Department of Psychiatry, Berlin